CLINICAL TRIAL: NCT00192517
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of MEDI-522, a Humanized Monoclonal Antibody to Integrin Alpha V Beta 3, Administered by Subcutaneous Injection to Adults With Plaque Psoriasis
Brief Title: Study of MEDI-522 Administered by Subcutaneous Injection to Adults With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Barbara White, M.D., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP102
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — etaracizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): MEDI-522
  Interventions: Drug: MEDI-522
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEDI-522 — 4 mg/kg (for 12 weeks based on patient's weight, to the nearest kg, obtained on Study Day 0)
  Arms: 1
Other: Placebo — 4 mg/kg(for 12 weeks based on patient's weight, to the nearest kg, obtained on Study Day 0)
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the effects on disease activity, in the absence of systemic psoriasis therapy, of 4 mg/kg MEDI-522 versus placebo administered weekly by SC injection for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis involving at least 10% of body surface area (Appendix A)
* PASI score greater than 12
* Age 18 through 65 years at the time of the first dose of study drug
* Both males and females are eligible. However, sexually active females, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 30 days prior to the first dose of study drug and must agree to continue using such precautions for 60 days after the final dose of study drug
* Prior to randomization (must be within 21 days of the first administration of the study drug), all of the following: WBC less than or equal to 3,800/mm3; hematocrit above 32%, platelet count less than or equal to 140,000/mm3; AST, ALT, BUN, or creatinine<1.5 x ULN; and stool negative for occult blood
* Currently receiving no therapy for psoriasis except emollients
* Written informed consent obtained from the patient
* Ability to complete follow-up period of 167 days as required by the protocol

Exclusion Criteria:

* Pustular, guttate, or erythrodermic psoriasis as the predominant disease type
* Evidence of active hepatitis A, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, such as positive HBsAg or positive anti-hepatitis C antibody
* Pregnancy (must have a negative serum pregnancy test within 21 days prior to the first dose of study drug, and urine pregnancy test must be negative on Study Day 0 before study entry)
* History of cancer (except excision of basal cell carcinoma)
* Evidence of significant active infection, such as fever less than or greater to 38.0°C (100.5°F), or chronic systemic infection
* Known or suspected infection with human immunodeficiency virus (HIV) or other evidence of clinically significant immune deficiencies
* Diagnosis of psoriatic arthritis or rheumatoid arthritis requiring active treatment
* History of hematuria due to chronic cystitis, recurrent kidney stones, or nephritis, history of CVA, poorly controlled hypertension, angina, stable abdominal aneurysm, recent superficial phlebitis, or recent myocardial infarction (within past 1 year without definitive corrective surgery such as coronary bypass graft or angioplasty)
* Receipt of systemic therapy for psoriasis or immunosuppressive medication in the past 4 weeks, including systemic retinoids, systemic steroids (oral, IM, or IV), cyclosporine A,methotrexate, azathioprine, anti-TNF agents, anti-T-cell agents, phototherapy (PUVA, UVB,tanning bed use), coal tar treatment (Goeckerman or modified Goeckerman regimen), tacrolimus, or mycophenolate
* Use of topical therapy for psoriasis in the past 2 weeks, such as steroid containing creams, Vitamin D analog creams and coal tar shampoos
* Receipt of any investigational drug therapy within 4 weeks before the first dose of study drug in this protocol (use of licensed agents for indications not listed in the package insert is permitted)
* Current or planned participation in a research protocol in which an investigational agent or therapy may be administered
* History of allergic disease or reactions likely to be exacerbated by any component of MEDI-522
* Nursing mother
* Evidence of acute illness
* Clinical manifestations of significant end organ dysfunction or failure that may compromise the safety of the patient in the study
* History of gastrointestinal bleeding (i.e., stool positive for occult blood or overt bleeding) within the previous 6 months
* Known bleeding disorder or significant risk of clinically important abnormal bleeding due to anticoagulant therapy with warfarin or heparin
* Insulin-dependent diabetes mellitus that is recent-onset or unstable
* Elective surgery planned during the study period through Study Day 167

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-12; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving at least a 50% or 75% improvement of PASI | PASI score at Study Days 28, 56, 77, 91, 107, 137, and 167.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | through Study Day 167

CONTACTS AND LOCATIONS:
Overall Officials: Barbara White, M.D., Study Director — MedImmune LLC
Locations (20):
- United States (18):
  - Bressinck, Gibson, Parker, Dinehart, Sanster Dermatology, PA, Little Rock, Arkansas
  - Associates In Research, Inc., Fresno, California
  - Solano Dermatology Associates, Vallejo, California
  - Dermatology Specialists, Vista, California
  - The Savin Center, P.C., New Haven, Connecticut
  - North Florida Dermatology Associates, P.A., Jacksonville, Florida
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - South Bend Clinic, South Bend, Indiana
  - FutureCare Studies, INC, Springfield, Massachusetts
  - Midwest Cutaneous Research, Corp., Clinton Township, Michigan
  - Central Dermatology, St Louis, Missouri
  - Karen Harkaway, M.D., LLC, Riverside Park, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - NorthEast Clinical Research Centers, Inc, Allentown, Pennsylvania
  - Clincial Partners, LLC, Johnston, Rhode Island
  - Harmony Clinical Research, Johnson City, Tennessee
  - Tenn. Clinical Research Center, INC, Nashville, Tennessee
  - Derm. Clinical Research Center of San Antonio, San Antonio, Texas
- Canada (2):
  - North Bay Dermatology Center, North Bay, Ontario
  - Probity Medical Research, Inc., Waterloo, Ontario